CLINICAL TRIAL: NCT03909295
Title: A Multicenter, Open-label Study to Evaluate the Safety and Tolerability of LCZ696 Treatment in Japanese Heart Failure Patients (NYHA Class II-IV) With Preserved Ejection Fraction After CLCZ696D2301 (PARAGON-HF)
Brief Title: An Open-label Extension Study Evaluating Safety and Tolerability of LCZ696 in Subjects Who Completed PARAGON-HF in Japan.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early because the primary endpoint of PARAGON-HF was not met.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696D1301E1
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Results first posted 2020-12-04 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFpEF)
Keywords: heart failure with preserved ejection fraction, Japanese patients, extension study, long-term safety and tolerability, open-label
MeSH Terms: interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCZ696 (Experimental): Starting dose was either 50 mg b.i.d. or 100 mg b.i.d. largely depending on the last dose level taken by the patient at the time of completing PARAGON-HF and patient condition. The dose level was gradually up-titrated with the goal of reaching the target dose of 200 mg b.i.d. as soon as tolerated by the patient
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696 — Starting dose was either 50 mg b.i.d. or 100 mg b.i.d. largely depending on the last dose level taken by the patient at the time of completing PARAGON-HF and patient condition. The dose level was gradually up-titrated with the goal of reaching the target dose of 200 mg b.i.d. as soon as tolerated by the patient
  Other Names: Sacubitril/valsartan

SUMMARY:
This study evaluated the safety and tolerability of LCZ696 treatment in Japanese heart failure patients (NYHA Class II-IV) with preserved ejection fraction after CLCZ696D2301 (PARAGON-HF).

DETAILED DESCRIPTION:
This study was an open-label extension study following the PARAGON-HF. Patients who have completed the PARAGON-HF were eligible to participate. During the study, open-label LCZ696 was taken in addition to background treatments of comorbidities. All subjects were treated with LCZ696 (sacubitril/valsartan) at maximally tolerated dosed with a target dose of 200 mg b.i.d (twice a day).

The subject were to continue to receive LCZ696 until it became commercially available, or for a period up to 24 months from the first patient enrolled in this study whichever came first. However, this study was terminated early based on the pre-defined early termination criteria of "the primary endpoint of PARAGONHF was not met" in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained before any assessment is performed.
* Patients who have completed LCZ696D2301 and are able to be safely enrolled into this study as judged by the investigator.

Exclusion Criteria:

* Patients who discontinued study drug treatment during LCZ696D2301 due to an event or intercurrent illness. Eligibility can be re-considered if the event has resolved and no longer represents a risk to the patient and the patient can safely tolerate the administration of LCZ696 per the investigator's assessment.
* Any medical condition that in the opinion of the investigator is likely to prevent the patient from safely tolerating LCZ696 or complying with the requirements of the study.
* Patients who have experience of angioedema event(s) which occurred and reported by the investigator during LCZ696D2301.
* Pregnant or nursing (lactating) women.
* Women of childbearing potential unless they are using highly effective methods of contraception.

Other protocol-defined inclusion/exclusion may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Japan (16):
  - Novartis Investigative Site, Seto, Aichi-ken
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Kan’onjichō, Kagawa-ken
  - Novartis Investigative Site, Takamatsu, Kagawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Sayama, Saitama
  - Novartis Investigative Site, Kusatsu, Shiga
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 52 participants were enrolled across 17 centers in Japan.
Pre-assignment Details: This study was terminated early based on the pre defined early termination criteria of "the primary endpoint of PARAGON-HF (CLCZ696D2301) was not met" in the protocol.
Period: Overall Study
Arm/Group | LCZ696
Started | 52
Safety Set (SAF) (All subjects who received at least one dose of study drug) | 52
Completed | 0
Not Completed | 52
Not completed — Adverse Event | 2
Not completed — Study terminated by sponsor | 50

BASELINE CHARACTERISTICS:
Arm/Group | LCZ696
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.37 (7.608)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a subject or clinical investigation subject after providing written informed consent for participation in the study. Any sign or symptom that occured from first dose of study treatment until end of study treatment.
Time Frame: Up to 27 weeks
Population: Safety set (SAF) included all participants who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- LCZ696 50 mg: Starting dose was either 50 mg b.i.d. or 100 mg b.i.d. largely depending on the last dose level taken by the patient at the time of completing PARAGON-HF and patient condition. The dose level was gradually up-titrated with the goal of reaching the target dose of 200 mg b.i.d. as soon as tolerated by the patient
Arm/Group | LCZ696 50 mg
Number analyzed (Participants) | 52
Participants
  Participants experiencing Adverse Events | 40
  Participants experiencing Serious Adverse Events | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment (up to 27 weeks).
Description: Any sign or symptom that occured from first dose of study treatment until end of study treatment (27 weeks).
Arm/Group | LCZ696
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 8/52
Other Adverse Events (participants affected / at risk) | 16/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=52)
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Macular fibrosis (Eye disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Embolic stroke (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 (N=52)
Diarrhoea (Gastrointestinal disorders) | 5
Nasopharyngitis (Infections and infestations) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03909295/Prot_001.pdf
  • Statistical Analysis Plan (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03909295/SAP_000.pdf